CLINICAL TRIAL: NCT05179187
Title: Non-invasive Brain Mapping of Movement Facilitation in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kathryn A. Cross, MD, PhD, Assistant Professor in Residence, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-002135; 1K23NS119568 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: movement; external cueing; brain mapping
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All participants undergo the same behavioral interventions in which upper extremity movements are made in response to different sensory stimuli.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson disease patients (Experimental): Participants diagnosed with Parkinson's disease
  Interventions: Behavioral: Movement task
- Healthy adults (Active Comparator): Healthy adult age-matched controls
  Interventions: Behavioral: Movement task

INTERVENTIONS:
Behavioral: Movement task — Computer task with experimental conditions manipulating sensory and motivation cues for movement.
  Other Names: Computer task

SUMMARY:
Several strategies or contexts help patients with Parkinson's disease to move more quickly or normally, however the brain mechanisms underlying these phenomena are poorly understood. The proposed studies use complimentary brain mapping techniques to understand the brain mechanisms supporting improved movements elicited by external cues. The central hypothesis is that distinct networks are involved in movement improvement depending on characteristics of the facilitating stimulus. Participants will perform movement tasks during recording of brain activity with EEG and MRI. The identified biomarkers may provide targets for future neuromodulation therapies to improve symptoms that are refractory to current treatments, such as freezing of gait.

DETAILED DESCRIPTION:
The studies proposed here test the overarching hypothesis that different types of cues (visual targets, rhythmic auditory stimuli and reward incentives) facilitate movement through distinct neuroanatomic circuits and electrophysiological mechanisms, by leveraging known variability in behavioral cueing benefits across patients.

Aim 1 is to demonstrate behavioral dissociations between different forms of movement facilitation within patients and relate variability in cueing benefits to integrity of dissociable neuroanatomic circuits as measured by resting state and diffusion tensor magnetic resonance imaging (MRI). Aim 2 is to characterize the electrophysiological correlates of behavioral benefits for the different cue types using electroencephalography (EEG).

Patients will perform two computer tasks involving reaching and tapping movements during video recording of movements and electrophysiological recording of brain signals. Experimental manipulations involve different computer stimuli that manipulate the presence or absence of sensory and motivational movement cues. The same experimental manipulations are delivered to all individual subjects. 60 patients with Parkinson's disease and 30 healthy controls will perform the task during recording of brain waves from the scalp (EEG) and return for a second session to record brain activity with MRI. Each of the total of 2 sessions will last about 1.5 hours. Patients may be asked to delay taking their morning Parkinson's disease medications and perform clinical rating scales and questionnaires and undergo a movement disorders neurological exam.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease based on presence of at least 2 cardinal features (tremor, rigidity or bradykinesia) OR healthy adult with no neurologic disease
* Age > 18 years old

Exclusion Criteria:

* Dementia as indicated by score on Montreal Cognitive Assessment < 19
* Active hallucinations or psychosis
* Contraindications to MRI (metal implant, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
EEG recordings | baseline
  EEG power in the beta band
BOLD fMRI: functional brain connectivity | up to 4 weeks
  Blood oxygen level dependent (BOLD) resting state network activity as a function of behavioral benefits from external cues
Diffusion tractography imaging (MRI): structural brain connectivity | up to 4 weeks
  Diffusion tensor fractional anisotropy as a function of behavioral benefits from external cues

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified resting state data and diffusion tractography (in raw form) will be available through the LONI Imaging and Data Archive (IDA) along with details of acquisition methods and clinical data and distributed upon approval by the PI. Electrophysiological and behavioral data obtained during task performance will be made available upon request to Dr. Cross (PI) via secured server access. Data sharing agreement will be required for all requests.